CLINICAL TRIAL: NCT06875752
Title: Is There a Need for Luteal Support in Modified Natural Cycle Frozen Embryo Transfer Cycles: a Prospective, Multicenter, Randomized Trial
Brief Title: Is There a Need for Luteal Support in Modified Natural Cycle Frozen Embryo Transfer Cycles
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dunamenti REK Istenhegyi IVF Center (Other)
Collaborators: Medical University of Pecs (Other); Dunamenti REK Gyor Clinic (Unknown); Dunementi REK Pannon Clinic (Unknown); University of Szeged, Hungary (Unknown)
Responsible Party: Principal Investigator, Peter Kovacs MD, medical director Dunamenti REK Istenhegyi IVF Center, Dunamenti REK Istenhegyi IVF Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NNGYK/16437-3/2025
Record Dates: First submitted 2025-03-05; First posted 2025-03-13 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Luteal Support; Frozen Embryo Transfer (FET)
Keywords: luteal support; frozen embryo transfer; progesterone; modified natural cycle
MeSH Terms: interventions — Progesterone; Utrogestan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- No luteal support during modified natural cycle frozen embryo transfer (Active Comparator): In this arm the patient has her first ultrasound scheduled between days 9-12 of the cycle; the scan is repeated in 2-3 days if the follicle is not large enough or if the endometrium is thin (<7 mm). Serum progesterone measurement at the time of the last ultrasound. If the progesterone level is <1.5 ng/ml and the follicle has reached at least 17 mm in diameters hCG (250 mcg recombinant hCG, Ovitrelle) is administered in the evening hours (7-10 PM) 5-6 days after the trigger injection, latest in the AM of the planned FET, serum progesterone is measured again. If the value is under 10 ng/ml (31.8 nmol/l) vaginal luteal support is initiated and while we will proceed with the ET, the patient drops out of the RCT. If the progesterone is >31.8 nmol/l the patient receives no luteal support in this arm. 7 days after the hCG trigger she proceeds with the frozen embryo transfer.
  Interventions: Drug: no luteal support
- Vaginal progesterone luteal support (Active Comparator): In this arm the patient has her first ultrasound scheduled between days 9-12 of the cycle; the scan is repeated in 2-3 days if the follicle is not large enough or if the endometrium is thin (<7 mm). Serum progesterone measurement at the time of the last ultrasound. If the progesterone level is <1.5 ng/ml and the follicle has reached at least 17 mm in diameters hCG (250 mcg recombinant hCG, Ovitrelle) is administered in the evening hours (7-10 PM) 5-6 days after the trigger injection, latest in the AM of the planned FET, serum progesterone is measured again. If the value is under 10 ng/ml (31.8 nmol/l) vaginal luteal support is initiated and while we will proceed with the ET, the patient drops out of the RCT. If the progesterone is >31.8 nmol/l the patient in this arm still receives additional 2x200 mg vaginal progesterone luteal support (Utrogestan) starting on the day of embryo trasfer. 7 days after the hCG trigger she proceeds with the frozen embryo transfer.
  Interventions: Drug: Vaginal Progesterone
- Vaginal progesterone plus small dose hCG luteal support (Active Comparator): In this arm the patient has her first ultrasound scheduled between days 9-12 of the cycle; the scan is repeated in 2-3 days if the follicle is not large enough or if the endometrium is thin (<7 mm). Serum progesterone measurement at the time of the last ultrasound. If the progesterone level is <1.5 ng/ml and the follicle has reached at least 17 mm in diameters hCG (250 mcg recombinant hCG, Ovitrelle) is administered in the evening hours.5-6 days after the trigger injection, serum progesterone is measured again. If the value is under 10 ng/ml (31.8 nmol/l) vaginal luteal support is initiated and while we will proceed with the ET, the patient drops out of the RCT. If the progesterone is >31.8 nmol/l the patient in this arm receives 2x200 mg vaginal progesterone luteal support (Utrogestan) starting on the day of ET + 125 mcg rHCG s.c. on the day of ET and 62.5 mcg rHCG s.c. 4 days later. 7 days after the hCG trigger she proceeds with the frozen embryo transfer.
  Interventions: Drug: Progesterone plus HCG

INTERVENTIONS:
Drug: no luteal support — In one arm of the study the patients receive no luteal support as part of their modified natural cycle frozen embryo transfer.
  Arms: No luteal support during modified natural cycle frozen embryo transfer
Drug: Vaginal Progesterone — In the 2nd arm the patient receives 2x200 mg vaginal progesterone as luteal support.
  Arms: Vaginal progesterone luteal support
Drug: Progesterone plus HCG — In the 3rd arm the patients receive 2x200 mg vaginal progesteroen plus 125 mcg recombinant HCG s.c. on the day of embryo transfer and 62.5 mcg recombinant HCG s.c. 4 days later.
  Other Names: Utrogestan
  Arms: Vaginal progesterone plus small dose hCG luteal support

SUMMARY:
Without progesterone there is no pregnancy. Following ovulation, the endocrine function of the follicle changes and progesterone replacing estradiol becomes its main secretory product. In the follicular phase the increasing amount of estradiol secreted by the growing follicle builds up the endometrium, while in the luteal phase progesterone, the main product of the corpus luteum, prepares the endometrium for implantation. This process is called decidualization. If implantation occurs, human chorionic gonadotropin (hCG) secreted by the trophopblasts maintains the function of the corpus luteum. This continued activity is required to be maintained up to week 7-9 of gestation when the hormone secreting activity is taken over by the placenta (luteo-placental shift) and the corpus luteum regresses.

During in vitro fertilization (IVF) gonadotropins are used to induce multifollicular development and therefore following the oocyte retrieval ("ovulation") multiple corpora lutea are formed. At the same time, partly due to the supraphysiologic steroid levels reached during stimulation and partly to the removal of the granulosa cell mass during the retrieval, the activity of these corpora lutea remains insufficient and luteal support, primarily in the form of progesterone, is needed to achieve success.

Embryo cryopreservation has become available soon after the first successful IVF treatment. In some of the IVF treatments cryopreservation is electively planned, while in others surplus embryos are frozen. As a result of the currently available vitrification technology a close to 100% survival can be expected upon thawing.

Frozen embryos can be transferred according to different protocols:

1. True natural cycle FET (tNC-FET): in these cases, spontaneous follicle growth is followed by spontaneous ovulation and the timing of the embryo transfer (ET) is timed according to the spontaneous luteinizing hormone (LH) surge
2. Modified natural cycle FET (mNC-FET): in these cases, follicle growth is spontaneous but ovulation is induced with hCG injection as soon as the follicle reaches maturity and the ET is timed to the trigger injection
3. Stimulated cycle FET (sNC-FET): in these cases, follicle growth is induced with oral agents or gonadotropins and once the lead follicle reaches maturity hCG injection is given to induce ovulation and the ET is timed to the trigger injection
4. Artificial, hormone replacement cycle (HRT-FET): in these cases, the ovaries are not active but estradiol is given to build up the endometrium and once proper thickness is reached progesterone is added to prepare to implantation According to the available evidence the different approaches are equally effective. The common theme in mNC, tNC and sNC FET cycles is that a corpus luteum is formed and its activity is not compromised by supraphysiologic steroid levels and the oocyte retrieval either. Despite this, in most clinics, similarly to the fresh IVF-ETs, luteal support is administered in FET cycles as well. The benefit of luteal support in NC-FET cycles is questionable, however. The available literature is inconclusive whether there is a need for luteal support in mNC-FET treatments? In order to answer this question, the investigators plan to perform a prospective, multicenter randomized pilot study.

Eligible participants will be randomized to one of the following groups:

1. No luteal support
2. 2x200 mg vaginal progesterone luteal support (Utrogestan) starting on the day of ET
3. 2x200 mg vaginal progesterone luteal support (Utrogestan) starting on the day of ET + 125 mcg rHCG s.c. (1/2 amp Ovitrelle) on the day of ET and 62.5 mcg rHCG s.c. (1/4 amp Ovitrelle) 4 days later.

Baseline demographic, FET treatment related, and clinical outcomes will be compared in the three different luteal phase management groups.

DETAILED DESCRIPTION:
Aim: The aim of this RCT is to assess whether the use of luteal support improves the outcome of modified natural cycle frozen embryo transfer (FET) treatments.

Background: Without progesterone there is no pregnancy. Following ovulation, the endocrine function of the follicle changes and progesterone replacing estradiol becomes its main secretory product. In the follicular phase the increasing amount of estradiol secreted by the growing follicle builds up the endometrium, while in the luteal phase progesterone, the main product of the corpus luteum, prepares the endometrium for implantation. This process is called decidualization. If implantation occurs, human chorionic gonadotropin (hCG) secreted by the trophopblasts maintains the function of the corpus luteum. This continued activity is required to be maintained up to week 7-9 of gestation when the hormone secreting activity is taken over by the placenta (luteo-placental shift) and the corpus luteum regresses.

During in vitro fertilization (IVF) gonadotropins are used to induce multifollicular development and therefore following the oocyte retrieval ("ovulation") multiple corpora lutea are formed. At the same time, partly due to the supraphysiologic steroid levels reached during stimulation and partly to the removal of the granulosa cell mass during the retrieval, the activity of these copora lutea remains insufficient and luteal support, primarily in the form of progesterone, is needed to achieve success.

Embryo cryopreservation has become available soon after the first successful IVF treatment. In some of the IVF treatments cryopreservation is electively planned, while in others surplus embryos are frozen. As a result of the currently available vitrification technology a close to 100% survival can be expected upon thawing.

Frozen embryos can be transferred according to different protocols:

1. True natural cycle FET (tNC-FET): in these cases, spontaneous follicle growth is followed by spontaneous ovulation and the timing of the embryo transfer (ET) is timed according to the spontaneous luteinizing hormone (LH) surge
2. Modified natural cycle FET (mNC-FET): in these cases, follicle growth is spontaneous but ovulation is induced with hCG injection as soon as the follicle reaches maturity and the ET is timed to the trigger injection
3. Stimulated cycle FET (sNC-FET): in these cases, follicle growth is induced with oral agents or gonadotropins and once the lead follicle reaches maturity hCG injection is given to induce ovulation and the ET is timed to the trigger injection
4. Artificial, hormone replacement cycle (HRT-FET): in these cases, the ovaries are not active but estradiol is given to build up the endometrium and once proper thickness is reached progesterone is added to prepare to implantation According to the available evidence the different approaches are equally effective. Many clinics favor the HRT cycle as it allows flexible scheduling of the embryo transfer. Recent publications have reported a higher incidence of hypertensive complications during pregnancies conceived in an HRT cycle though. This observation shifted to focus again on the natural cycle FET treatments.

The common theme in mNC, tNC and sNC FET cycles is that a corpus luteum is formed and its activity is not compromised by supraphysiologic steroid levels and the oocyte retrieval either. Despite this, in most clinics, similarly to the fresh IVF-ETs, luteal support is administered in FET cycles as well. The benefit of luteal support in NC-FET cycles is questionable, however. Various groups have studied the potential advantages of luteal support in the different types on NC-FET cycles.

One study has shown that the chance of live birth was reduced (25.7% vs 41.1%) in tNC FET cycles when the serum progesterone level was below 10 ng/ml. Another study, based on the outcome of close to 400 FET cycles, failed to find a benefit with luteal support. Based on the outcome of different types of FET cycles however, they observed a lower live birth rate when the serum progesterone level was below 7.8 ng/ml. Finally, they also observed suboptimal outcome when the serum progesterone level was over 20.3 ng/ml. Finally, a different group, did not find a difference in the progesterone levels among pregnant and non-pregnant participants not using luteal support in an RCT. They were also unable to identify a progesterone level that could discriminate among pregnant and non-pregnant women.

Several RCTs evaluated the potential benefits of luteal support. One research group has randomly assigned women to luteal support vs no luteal support in an RCT of mNC-FET. Clinical pregnancy, miscarriage and live birth rates were similar in the two groups. Another group, in a study of similar design also failed to show improved clinical outcome with luteal support in mNC-FET cycles. Two larger RCTs of tNC-FET however have reported improved clinical outcome with luteal support. Meta-analyses have reported conflicting results. One has shown improved live birth rate with luteal support in tNC-FET while found no benefit in mNC-FET cycles. Whiel two other meta-analyses have found higher clinical pregnancy rates in cycles with progesterone support. In summary, one can conclude that the literature is conflicting on the benefits of luteal support in mNC-FET cycles and even discuss a potential negative effect of high serum progesterone levels.

Based on the above the question arises whether there is a need for luteal support in mNC-FET treatments? Study protocol: In order to answer this question, the investigators plan to perform a prospective, multicenter randomized pilot study.

The investigators plan to enroll women between the ages of 18-40 (at the time of vitrification) who have at least one good morphology blastocyst (BC) frozen (morphology 2AA, 2AB, 2BA, 2BB, 3AA, 3AB, 3BA, 3BB, 4AA, 4AB, 4BA, 4BB, 5AA, 5AB, 5BA, 5BB using the Gardner classification) and who plan to undergo single frozen-thawed blastocyst transfer. In addition, the following inclusion criteria apply:

* Age 18-40 years at the time of vitrification
* At least one good quality BC frozen
* Planned 1 BC ET
* < 3 failed previous ETs
* Cycle length between 21-35 days
* Body mass index (BMI): 18-35 kg/m2
* Intact uterine cavity based on hysteroscopy, hysteron-salpingogram, salina sonohysterogram
* Consent to participate

The following exclusion criteria will apply:

* Age <18 of over 40 at the time of vitrification
* BMI: <18 kg/m2 or >35 kg/m2
* Planned ET of more than 1 embryo
* Irregular cycles (<21 or >35 days)
* Use of a protocol other than the mNC-FET
* Lack of good morphology blastocysts
* No evidence for spontaneous follicle development (no dominant (>17 mm) follicle by day 20 of cycle)
* Patient with a history of recurrent miscarriages
* Presence of a hydrosalpinx
* Irregular uterine cavity
* Positive test for HIV, hepatitis B or C
* Lack of consent
* Contraindication to the use of hCG or vaginal progesterone
* Use of blood thinners (aspirin, low molecular weight heparin)

Treatment protocol:

* Prior to the start of the FET cycle (latest at the first folliculometry) informed consent is obtained
* A first ultrasound is scheduled between days 9-12 of the cycle; the scan is repeated in 2-3 days if the follicle is not large enough or if the endometrium is thin (<7 mm)
* Serum progesterone measurement at the time of the last ultrasound. If the value is >1.5 ng/ml, the cycle is cancelled. If the progesterone level is <1.5 ng/ml and the follicle has reached at least 17 mm in diameters hCG (250 mcg recombinant hCG, Ovitrelle) is administered in the evening hours (7-10 PM)
* 5-6 days after the trigger injection, latest in the AM of the planned FET, serum progesterone is measured again. If the value is under 10 ng/ml (31.8 nmol/l) vaginal luteal support is initiated and while we will proceed with the ET, the patient drops out of the RCT. In these cases, the investigators apply "progesterone rescue" as it has been shown to maintain clinical efficacy when the progesterone levels is low before the transfer.
* Those who have a progesterone level >10 ng/ml (31.8 nmol/l) will be randomized to one of the following 3 groups on the day of FET (rHCG + 7):

  1. No luteal support
  2. 2x200 mg vaginal progesterone luteal support (Utrogestan) starting on the day of ET
  3. 2x200 mg vaginal progesterone luteal support (Utrogestan) starting on the day of ET + 125 mcg rHCG s.c. (1/2 amp Ovitrelle) on the day of ET and 62.5 mcg rHCG s.c. (1/4 amp Ovitrelle) 4 days later. Based on very limited data a potential negative effect of high luteal phase progesterone level was raised. It can be presumed that high progesterone, via negative feed-back, lowers pituitary LH release and may cause luteal insufficiency and ultimately could be responsible for reduced clinical success. Should this be the case, the additional small doses of hCG administered on the day of ET and 4 days later could "rescue" the corpus luteum. This is the rational for additional hCG use in the 3rd group.
* 6-8 days after the ET serum progesterone will be measured
* 12-13 days after the ET serum beta hCG and progesterone will be measured to check for implantation
* 3 +/- 0.5 weeks later vaginal ultrasound will be performed to check for clinical pregnancy
* Repeat ultrasound will be done at week 10-12 of gestation (by the primary obstetrician provider) to assess for ongoing pregnancy
* At the completion of pregnancy data will be collected on outcome parameters (potential hypertensive complications [gestational hypertension, pre-eclampsia, eclampsia] during pregnancy, gestational age at delivery, birthweight, APGAR score) Randomization: randomization will be made according to a computer-generated randomization list (www.randomizer.org). The prepared list will be accessible to all sub-investigators online. Participants who sign an informed consent and reach the trigger hCG injection will be assigned the next treatment option on the randomization list.

Blinding: neither the participants, nor the investigators will be blinded for assignment.

Placebo: the study will not involve the use of placebo. Drop-out: Participants who do not reach the hCG trigger day despite signing a consent form drop out of the study (true dropouts) and will not be randomized. Those who are randomized but do not have an ET for no available embryo to transfer after thawing, or other reasons will be kept in the intent-to-treat analysis but will not be considered in the per protocol analysis.

Sample size calculation: Since it is not known what the expected pregnancy rate without luteal support would be and whether that would be any different compared to treatments involving luteal support as a first step, the investigators plan a pilot study. The goal is to have 180 patients sign informed consent (60 potential patients per arm). 20% of the participants are expected not to reach the ET (lack of follicle development, other complications prior to the day of ET, no available embryos after thawing) that would leave the study with 150 patients treated per protocol.

Data collection: Data will be collected in structured Excel files. No patient identifying parameter (name, ID number) will be included just the randomization number. The name associated with the randomization number will be collected in a separate file by the sub investigator and will not be forwarded to the principal investigator. The principal investigator will only receive the anonymized data, and the combined anonymous dataset will be shared with the statistician. The following parameters will be collected:

* Age at cryopreservation
* Number of previous ETs
* BMI
* Smoking (yes-no)
* Progesterone level prior to trigger (nmol/l)
* Day of trigger calculation from day 1 of cycle
* Endometrial thickness at the last scan (mm)
* Exact embryo quality (Gardner score)
* Ease of ET (two categories: easy vs difficult [need for tenaculum, sedation, stiff catheter])
* Progesterone level 6-8 days after rHCG trigger
* HCG and progesterone 12-13 days after ET
* Clinical pregnancy (intrauterine gestational sac; yes-no)
* Ongoing, live pregnancy at week 10-12 (yes-no)
* Live birth
* Miscarriage (early: before week 12; late week 12-24.)
* Single vs multiple pregnancy
* Gestational age at delivery
* Vaginal vs Cesarean delivery
* Birth weight
* APGAR score
* Hypertensive complication during pregnancy (yes vs no)

Definitions:

* Biochemical pregnancy: hCG>10 IU/l
* Clinical pregnancy: intrauterine gestational sac
* Ongoing pregnancy: embryo with heartbeat at week 10-12
* Early miscarriage: pregnancy loss prior to week 12
* Late miscarriage: pregnancy loss week 12-24
* Live birth: delivery after 24 weeks gestation
* Preterm delivery: deliver prior to week 37 gestation
* Very preterm delivery: delivery before week 32 gestation
* Low birth weight: < 2500 g
* Very low birth weight: < 1500 g

Statistical analysis: Baseline demographic, FET treatment related, and clinical outcomes will be compared in the three different luteal phase management groups. Continuous variables will be shown as mean +/- SD, while categorical variable as number and percent. ANOVA and Mann-Whitney U test will be used for the analysis. Subgroups analysis is planned based on progesterone levels both prior to the trigger (31.8-50, 50-100, >100 nmol/l.) and 6-8 days after the trigger (< 31.8, 31.8-50, 50-100, >100 nmol/l). analysis will be performed based on intent-to-treat and per protocol as well. Post hoc comparison of the different treatment groups to each other will be performed.

References:

1. Csapo AI, Pulkkinen MO, Wiest WG.Effects of luteectomy and progesterone replacement therapy in early pregnant patients. Am J Obstet Gynecol. 1973 Mar 15;115(6):759-65. doi: 10.1016/0002-9378(73)90517-6.
2. Trounson A, Mohr L. Human pregnancy following cryopreservation, thawing and transfer of an eight-cell embryo. Nature. 1983 Oct 20-26;305(5936):707-9. doi: 10.1038/305707a0.)
3. Lawrenz B, Coughlan C, Melado L, Fatemi HM. The ART of frozen embryo transfer: back to nature! Gynecol Endocrinol. 2020 Jun;36(6):479-483. doi: 10.1080/09513590.2020.1740918.
4. Glujovsky, R Pesce, C Sueldo, AMQ Retamar, RJ Hart, A Ciapponi. Endometrial preparation for women undergoing embryo transfer with frozen embryos or embryos derived from donor oocytes. Cochrane Database Syst Rev 2020 Oct 28;10(10):CD006359.
5. Bortoletto P, Prabhu M, Baker VL. Association between programmed frozen embryo transfer and hypertensive disorders of pregnancy. Fertil Steril. 2022 Nov;118(5):839-848. doi: 10.1016/j.fertnstert.2022.07.025.
6. Gaggiotti-Marre S, Álvarez M, González-Foruria I, Parriego M, Garcia S, Martínez F, Barri PN, Polyzos NP, Coroleu B. Low progesterone levels on the day before natural cycle frozen embryotransfer are negatively associated with live birth rates. Hum Reprod. 2020 Jul 1;35(7):1623-1629. doi: 10.1093/humrep/deaa092.
7. Melo P, Wood S, Petsas G, Chung Y, Easter C, Price MJ, Fishel S, Khairy M, Kingsland C, Lowe P, Rajkhowa M, Sephton V, Pandey S, Kazem R, Walker D, Gorodeckaja J, Wilcox M, Gallos I, Tozer A, Coomarasamy A. The effect of frozen embryo transfer regimen on the association between serum progesterone and live birth: a multicentre prospective cohort study (ProFET). Hum Reprod Open. 2022 Nov 28;2022(4):hoac054. doi: 10.1093/hropen/hoac054.
8. Saupstad M, Bergenheim SJ, Bogstad JW, Petersen MR, Klajnbard A, Prætorius L, Freiesleben NLC, Englund AL, Løkkegaard ECL, Knudsen UB, Husth M, Alsbjerg B, Møller JE, Dam TV, Forman JL, Pinborg A, Løssl K. Progesterone concentrations on blastocyst transfer day in modified natural cycle frozen embryo transfer cycles. Reprod Biomed Online. 2024 Jul;49(1):103862. doi: 10.1016/j.rbmo.2024.103862.
9. Horowitz E, Mizrachi Y, Finkelstein M, Farhi J, Shalev A, Gold E, Raziel A, Weissman A. A randomized controlled trial of vaginal progesterone for luteal phase support in modified natural cycle - frozen embryo transfer. Gynecol Endocrinol. 2021 Sep;37(9):792-797. doi: 10.1080/09513590.2020.1854717.
10. Eftekhar M, Rahsepar M, Rahmani E. Effect of progesterone supplementation on natural frozen-thawed embryotransfer cycles: a randomized controlled trial. Int J Fertil Steril. 2013 Apr;7(1):13-20.
11. Wånggren K, Dahlgren Granbom M, Iliadis SI, Gudmundsson J, Stavreus-Evers A. Progesterone supplementation in natural cycles improves live birth rates after embryo transfer of frozen-thawed embryos-a randomized controlled trial. Hum Reprod. 2022 Sep 30;37(10):2366-2374. doi: 10.1093/humrep/deac181.
12. Kerstin Bjuresten, Britt-Marie Landgren, Outi Hovatta, Anneli Stavreus-Evers. Luteal phase progesterone increases live birth rate after frozen embryo transfer. Fertil Steril 2011 Feb;95(2):534-7.doi: 10.1016/j.fertnstert.2010.05.019.
13. Jiang Y, Wang L, Shen H, Wang B, Wu J, Hu K, Wang Y, Ma B, Zhang X. The effect of progesterone supplementation for luteal phase support in natural cycle frozen embryo transfer: a systematic review and meta-analysis based on randomized controlled trials. Fertil Steril. 2023 Apr;119(4):597-605. doi: 10.1016/j.fertnstert.2022.12.035.
14. Mizrachi Y, Horowitz E, Ganer Herman H, Farhi J, Raziel A, Weissman A. Should women receive luteal support following natural cycle frozen embryotransfer? A systematic review and meta-analysis. Hum Reprod Update. 2021 Jun 22;27(4):643-650. doi: 10.1093/humupd/dmab011.
15. Su S, Zeng M, Duan J. Luteal phase support for natural cycle frozen embryo transfer: a meta-analysis. Gynecol Endocrinol. 2022 Feb;38(2):116-123. doi: 10.1080/09513590.2021.1998438.
16. Gardner DK, Sakkas D. Assessment of embryo viability: the ability to select a single embryo for transfer - a review. Placenta 2003;24, Suppl. B:S5-12.
17. Stavridis K, Kastora SL, Triantafyllidou O, Mavrelos D, Vlahos N. Effectiveness of progesterone rescue in women presenting low circulating progesterone levels around the day of embryo transfer: a systematic review and meta-analysis. Fertil Steril. 2023 Jun;119(6):954-963. doi: 10.1016/j.fertnstert.2023.02.007.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years at the time of vitrification
* At least one good quality blastocyst frozen
* Planned 1 blastocyst transfer
* <3 failed previous ETs
* Cycle length between 21-35 days
* Body mass index (BMI): 18-35 kg/m2
* Intact uterine cavity based on hysteroscopy, hysteron-salpingogram, salina sonohysterogram
* Consent to participate

Exclusion Criteria:

* Age <18 of over 40 at the time of vitrification
* BMI: <18 kg/m2 or >35 kg/m2
* Planned transfer of more than 1 embryo
* Irregular cycles (<21 or >35 days)
* Use of a protocol other than the modified natural cycle frozen embryo transfer
* Lack of good morphology blastocysts
* No evidence for spontaneous follicle development (no dominant (>17 mm) follicle by day 20 of cycle)
* Patient with a history of recurrent miscarriages
* Presence of a hydrosalpinx
* Irregular uterine cavity
* Positive test for HIV, hepatitis B or C
* Lack of consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-04-12 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
ongoing clinical pregnancy | up to 3 months after the embryo transfer; starting with the first patient who has a positive pregnancy test after the frozen embryo transfer and up to 3 months after the completion of the study (last frozen embryo transfer)i.e.: last embryo transfer
  live intrauterine pregnancy at week 9-12 of gestation

CONTACTS AND LOCATIONS:
Locations (5):
- Hungary (5):
  - Dunamenti REK Istenhegyi IVF Center, Budapest, Budapest
  - Dunamenti REK Gyor IVF Center, Győr, Gyor
  - University of Pecs, Dept. OBGYN, Reproductive Center, Pécs, Pecs
  - University of Szeged, Reproductive Medicine Institute, Szeged, Szeged
  - Dunamenti REK Tapolca IVF Center, Tapolca, Tapolca

IPD SHARING:
Plan to Share IPD: Undecided
Patient data will be shared upon reasonable request.

REFERENCES:
- [Background] Stavridis K, Kastora SL, Triantafyllidou O, Mavrelos D, Vlahos N. Effectiveness of progesterone rescue in women presenting low circulating progesterone levels around the day of embryo transfer: a systematic review and meta-analysis. Fertil Steril. 2023 Jun;119(6):954-963. doi: 10.1016/j.fertnstert.2023.02.007. Epub 2023 Feb 11. PMID 36781098
- [Background] Su S, Zeng M, Duan J. Luteal phase support for natural cycle frozen embryo transfer: a meta-analysis. Gynecol Endocrinol. 2022 Feb;38(2):116-123. doi: 10.1080/09513590.2021.1998438. Epub 2021 Nov 3. PMID 34730071
- [Background] Jiang Y, Wang L, Shen H, Wang B, Wu J, Hu K, Wang Y, Ma B, Zhang X. The effect of progesterone supplementation for luteal phase support in natural cycle frozen embryo transfer: a systematic review and meta-analysis based on randomized controlled trials. Fertil Steril. 2023 Apr;119(4):597-605. doi: 10.1016/j.fertnstert.2022.12.035. Epub 2022 Dec 24. PMID 36574915
- [Background] Mizrachi Y, Horowitz E, Ganer Herman H, Farhi J, Raziel A, Weissman A. Should women receive luteal support following natural cycle frozen embryo transfer? A systematic review and meta-analysis. Hum Reprod Update. 2021 Jun 22;27(4):643-650. doi: 10.1093/humupd/dmab011. PMID 33829269
- [Background] Bjuresten K, Landgren BM, Hovatta O, Stavreus-Evers A. Luteal phase progesterone increases live birth rate after frozen embryo transfer. Fertil Steril. 2011 Feb;95(2):534-7. doi: 10.1016/j.fertnstert.2010.05.019. Epub 2010 Jun 26. PMID 20579989
- [Background] Wanggren K, Dahlgren Granbom M, Iliadis SI, Gudmundsson J, Stavreus-Evers A. Progesterone supplementation in natural cycles improves live birth rates after embryo transfer of frozen-thawed embryos-a randomized controlled trial. Hum Reprod. 2022 Sep 30;37(10):2366-2374. doi: 10.1093/humrep/deac181. PMID 35972453
- [Background] Horowitz E, Mizrachi Y, Finkelstein M, Farhi J, Shalev A, Gold E, Raziel A, Weissman A. A randomized controlled trial of vaginal progesterone for luteal phase support in modified natural cycle - frozen embryo transfer. Gynecol Endocrinol. 2021 Sep;37(9):792-797. doi: 10.1080/09513590.2020.1854717. Epub 2020 Dec 14. PMID 33307906
- [Background] Saupstad M, Bergenheim SJ, Bogstad JW, Petersen MR, Klajnbard A, Praetorius L, Freiesleben NLC, Englund AL, Lokkegaard ECL, Knudsen UB, Husth M, Alsbjerg B, Moller JE, Dam TV, Forman JL, Pinborg A, Lossl K. Progesterone concentrations on blastocyst transfer day in modified natural cycle frozen embryo transfer cycles. Reprod Biomed Online. 2024 Jul;49(1):103862. doi: 10.1016/j.rbmo.2024.103862. Epub 2024 Feb 6. PMID 38735231
- [Background] Melo P, Wood S, Petsas G, Chung Y, Easter C, Price MJ, Fishel S, Khairy M, Kingsland C, Lowe P, Rajkhowa M, Sephton V, Pandey S, Kazem R, Walker D, Gorodeckaja J, Wilcox M, Gallos I, Tozer A, Coomarasamy A. The effect of frozen embryo transfer regimen on the association between serum progesterone and live birth: a multicentre prospective cohort study (ProFET). Hum Reprod Open. 2022 Nov 28;2022(4):hoac054. doi: 10.1093/hropen/hoac054. eCollection 2022. PMID 36518987
- [Background] Gaggiotti-Marre S, Alvarez M, Gonzalez-Foruria I, Parriego M, Garcia S, Martinez F, Barri PN, Polyzos NP, Coroleu B. Low progesterone levels on the day before natural cycle frozen embryo transfer are negatively associated with live birth rates. Hum Reprod. 2020 Jul 1;35(7):1623-1629. doi: 10.1093/humrep/deaa092. PMID 32478389
- [Background] Bortoletto P, Prabhu M, Baker VL. Association between programmed frozen embryo transfer and hypertensive disorders of pregnancy. Fertil Steril. 2022 Nov;118(5):839-848. doi: 10.1016/j.fertnstert.2022.07.025. Epub 2022 Sep 25. PMID 36171152
- [Background] Glujovsky D, Pesce R, Sueldo C, Quinteiro Retamar AM, Hart RJ, Ciapponi A. Endometrial preparation for women undergoing embryo transfer with frozen embryos or embryos derived from donor oocytes. Cochrane Database Syst Rev. 2020 Oct 28;10(10):CD006359. doi: 10.1002/14651858.CD006359.pub3. PMID 33112418
- [Background] Lawrenz B, Coughlan C, Melado L, Fatemi HM. The ART of frozen embryo transfer: back to nature! Gynecol Endocrinol. 2020 Jun;36(6):479-483. doi: 10.1080/09513590.2020.1740918. Epub 2020 Mar 18. PMID 32188299
- [Background] Trounson A, Mohr L. Human pregnancy following cryopreservation, thawing and transfer of an eight-cell embryo. Nature. 1983 Oct 20-26;305(5936):707-9. doi: 10.1038/305707a0. PMID 6633637
- [Background] Csapo AI, Pulkkinen MO, Wiest WG. Effects of luteectomy and progesterone replacement therapy in early pregnant patients. Am J Obstet Gynecol. 1973 Mar 15;115(6):759-65. doi: 10.1016/0002-9378(73)90517-6. No abstract available. PMID 4688578